CLINICAL TRIAL: NCT03145311
Title: First Repetitive Transcranial Magnetic Stimulation for Treatment of Drug Induced Tardive Syndromes. Double Randomized Clinical Trial
Brief Title: First rTMS for Treatment of Drug Induced Tardive Syndromes. Double Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman M. Khedr, Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: rTMS in ttt of DITS
Record Dates: First submitted 2017-04-28; First posted 2017-05-09 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Drug Induced Tardive Syndrome (DITS)
Keywords: rTMS, Drug Induced Tardive Syndrome
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real rTMS (Active Comparator): Each patient received real repititive transcranial magnetic stimulation (rTMS) 20 HZ at 100% RMT (a total of 2000 pulses to each hand area consisting of 10 trains of 200 pulses with intertrain interval 30 s), over the hand motor area area for 10 consecutive days
  Interventions: Procedure: Repetitive transcranial magnetic stimulation (rTMS)
- Sham rTMS (Sham Comparator): Each patient received repetitive transcranial magnetic stimulation (rTMS) with the same pulse delivery as the 1st group but with the coil placed perpendicular to the scalp.
  Interventions: Procedure: Repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Procedure: Repetitive transcranial magnetic stimulation (rTMS)

SUMMARY:
This study aims to evaluate the efficacy of rTMS on DITS. Twenty patients with DITS were recruited from the outpatient clinic of Aswan University Hospital. The patients were classified into two equal groups, 1st group received real high frequency rTMS at 100% RMT and the 2nd group received sham stimulation with the same pulse delivery but with the coil placed perpendicular to the scalp. For each patient 10 sessions were administered once per day for 5 consecutive days each week for two weeks. All patients were assessed before rTMS and immediately after the end of the 10 sessions. This study is double blinded (the doctor and the patients). Assessment with AIMS scale and different parameters of cortical excitability were performed before and after the end of sessions treatment.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the efficacy of repetitive transcranial magnetic stimulation (rTMS) on drug induced tardive syndromes.

the effect of rTMS compare. Twenty patients with drug induced tardive syndromes were recruited from the outpatient clinic of Aswan University Hospital. The patients were classified into two equal groups, 1st group received real 20 Hz-rTMS at 100% RMT (a total of 2000 pulses to each hand area consisting of 10 trains of 200 pulses with intertrain interval 30 s), and the 2nd group received sham stimulation with the same pulse delivery as the 1st group but with the coil placed perpendicular to the scalp. For each patient 10 sessions were administered once per day for 5 consecutive days each week for two weeks. All patients were assessed before rTMS and immediately after the end of the 10 sessions. The patients did not know which type of stimulation they received and to ensure that, the study was double blinded the doctor who assessed the patients didn't know which type of stimulation the patients received. None of the patients had had rTMS before and were unaware of the type of stimulation.The AIMS scale and different parameters of cortical excitability were assessed before and after the end of session treatment.

ELIGIBILITY:
Inclusion Criteria:

* All patients with the spectrum of Tardive dyskinesia (TD) according to the diagnostic and statistical manual of mental disorders, fourth edition (DSM IV)

Exclusion Criteria:

* None of the patients suffered from any other clinically relevant disorders.
* We exclude any patient with pacemaker or metallic devices
* patients with history of epilepsy or metabolic diseases.

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Change in AIMS score | An average one month
  Measure the change in AIMS score at the end of the 10th session and then one month later.

SECONDARY OUTCOMES:
Changes in cortical excitability | 10 days
  Measure the change in cortical excitability before the 1st and then after the 10th session

CONTACTS AND LOCATIONS:
Overall Officials: Eman M Khedr, MD, Principal Investigator — Professor of Neurology, Faculty of Medicine, Assiut University
Locations (1):
- Eman Khedr, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khedr EM, Al Fawal B, Abdelwarith A, Saber M, Rothwell JC. Repetitive transcranial magnetic stimulation for treatment of tardive syndromes: double randomized clinical trial. J Neural Transm (Vienna). 2019 Feb;126(2):183-191. doi: 10.1007/s00702-018-1941-x. Epub 2018 Oct 13. PMID 30317532